CLINICAL TRIAL: NCT03871036
Title: ICRA (Improve Checkpoint-blockade Response in Advanced Urothelial Cancer), an Adaptive Clinical Study to Determine Efficacy of Combining Weekly Paclitaxel With Tremelimumab +/- Durvalumab (MEDI4736)
Brief Title: Improve Checkpoint-blockade Response in Advanced Urothelial Cancer
Acronym: ICRA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M18ICR/ESR-18-13667
Record Dates: First submitted 2019-02-14; First posted 2019-03-12 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma
Keywords: Advanced urothelial carcinoma; Checkpoint inhibition; Tremelimumab; Durvalumab; Paclitaxel
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — tremelimumab; durvalumab; Paclitaxel

STUDY DESIGN:
Intervention Model Description: A run-in safety phase will be followed by a non-comparative 3-arm randomized study with a Simon's 2-stage optimal design. Run-in safety phase will start with an increasing dose of tremelimumab in combination with paclitaxel. In the final part of the run-in safety phase, patients will be randomized to receive paclitaxel with either regular dose tremelimumab in combination with durvalumab, or a high dose tremelimumab. If no unexpected toxicity occurs, the experimental phase of the study will start, randomizing patients over 3 arms. The best arm will be expanded based on a Simon's 2-stage optimal design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Tremelimumab 75 (R1) (Experimental): Run-in phase-1 (R1): n=3 patients will be treated with:
  * paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
  * tremelimumab 75 mg on day 1 of cycles 2-6 and then every 12 weeks until week 45
  Interventions: Drug: Tremelimumab; Drug: Paclitaxel
- Tremelimumab 225 (R2) (Experimental): Run-in phase-2 (R2): n=3 patients will be treated with:
  * paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
  * tremelimumab 225 mg on day 1 of cycles 2-6 and then every 12 weeks until week 45
  Interventions: Drug: Tremelimumab; Drug: Paclitaxel
- Tremelimumab vs Tremelimumab+Durvalumab (R3) (Experimental): Run-in phase-3 (R3): n=2 x 3 patients will be randomized over 2 arms:
  * paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
  * tremelimumab 750 mg on day 1 of cycles 2-6 and then every 12 weeks until week 45
  OR
  * paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
  * tremelimumab 75 mg on day 1 of cycles 2-5
  * durvalumab 1500 mg on day 1 of cycles 2-12, every four weeks (until week 49)
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Drug: Paclitaxel
- Tremelimumab 300 (R4) (Experimental): Run-in phase-4 (R4): n=3 patients will be treated with:
  * paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
  * tremelimumab 300 mg once on day 1 of cycle 2
  * durvalumab 1500 mg on day 1 of cycles 2-12, every four weeks (until week 49)
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Drug: Paclitaxel
- Tremelimumab 750 (A) (Experimental): Arm A:
  * paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
  * tremelimumab 750 mg on day 1 of cycles 2-6 and then every 12 weeks until week 45
  Interventions: Drug: Tremelimumab; Drug: Paclitaxel
- Tremelimumab+Durvalumab (B) (Experimental): Arm B:
  * paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
  * tremelimumab 300 mg once on day 1 of cycle 2
  * durvalumab 1500 mg on day 1 of cycles 2-12, every four weeks (until week 49)
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Drug: Paclitaxel
- Tremelimumab without paclitaxel (C) (Experimental): Arm C (control arm):
  • tremelimumab 750 mg on day 1 of cycles 1-5 and then every 12 weeks until week 41
  Interventions: Drug: Tremelimumab

INTERVENTIONS:
Drug: Tremelimumab — See experimental arm description for more details.
  Other Names: Ticilimumab; CP-675,206
Drug: Durvalumab — See experimental arm description for more details.
  Other Names: Imfinzi; MEDI4736
  Arms: Tremelimumab 300 (R4); Tremelimumab vs Tremelimumab+Durvalumab (R3); Tremelimumab+Durvalumab (B)
Drug: Paclitaxel — See experimental arm description for more details.
  Other Names: Taxol
  Arms: Tremelimumab 225 (R2); Tremelimumab 300 (R4); Tremelimumab 75 (R1); Tremelimumab 750 (A); Tremelimumab vs Tremelimumab+Durvalumab (R3); Tremelimumab+Durvalumab (B)

SUMMARY:
This trial will include metastatic urothelial carcinoma patients who progressed during or after treatment with anti-PD(L)1 therapy and have been treated by a platinum-containing regimen, or are cisplatin-ineligible. Patients will receive either paclitaxel in combination with durvalumab (anti-PDL-1) and a single dose (300 mg) of tremelimumab (anti-CTLA4), or paclitaxel with only a high dose of tremelimumab (750 mg). Tremelimumab (750 mg), without paclitaxel will be used as a comparison arm.

A run-in safety phase will be followed by a non-comparative 3-arm randomized study with a Simon's 2-stage optimal design.

DETAILED DESCRIPTION:
This trial will include metastatic urothelial carcinoma patients who progressed during or after treatment with anti-PD(L)1 therapy and have been treated by a platinum-containing regimen, or are cisplatin-ineligible.

A run-in safety phase will be followed by a non-comparative 3-arm randomized study with a Simon's 2-stage optimal design.

Screening:

Before enrollment, patients will need to complete the following screening procedures (among other assessments):

* Baseline evaluation by CT chest/abdomen/pelvis (<4 weeks)
* Laboratory assessment
* Tissue biopsy (in at least 6 patients per arm)

Run-in phase-1 (R1): n=3 patients will be treated with:

* paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
* tremelimumab 75 mg on day 1 of cycles 2-6 and then every 12 weeks until week 45

Run-in phase-2 (R2): n=3 patients will be treated with:

* paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
* tremelimumab 225 mg on day 1 of cycles 2-6 and then every 12 weeks until week 45

Run-in phase-3 (R3): n=2 x 3 patients will be randomized over 2 arms:

* paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
* tremelimumab 750 mg on day 1 of cycles 2-6 and then every 12 weeks until week 45 OR
* paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
* tremelimumab 75 mg on day 1 of cycles 2-5
* durvalumab 1500 mg on day 1 of cycles 2-12, every four weeks (until week 49)

Run-in phase-4 (R4): n=3 patients will be treated with:

* paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
* tremelimumab 300 mg once on day 1 of cycle 2
* durvalumab 1500 mg on day 1 of cycles 2-12, every four weeks (until week 49)

Enrollment will start with the first run-in cohort (R1) and will be halted after inclusion of the 3rd patient, until 60 days after start of treatment of this patient. Stopping rules are defined in the section 6.3 of the protocol. In case unexpected toxicity occurs (either as defined by the stopping rules or otherwise unexpected severe toxicity), the study team will discuss with the IDMC whether expansion to include 3 additional subjects is warranted. If no unexpected toxicity has occurred within 60 days after initiation of treatment of the 3rd patient of R1, enrollment for R2 will begin in a similar fashion. If 2 or more nonhematological toxicities as described in section 6.3 "Definition of DLT" occur in R1 or R2, enrollment will be suspended until the IDMC has formulated an advice. After this advice, the sponsor will decide on continuation.

If no unexpected toxicity has occurred within 60 days after initiation of treatment of the 3rd patient of R2, the study will continue with a third run-in cohort (R3) where patients will be randomized over 2 arms (R3A and R3B), n=3 per arm. If no unexpected toxicity has occurred within 60 days after initiation of treatment of the 3rd patient in arm R3A, this arm will be continued into the main study phase (as Arm A). If unacceptable toxicity is observed at either 225 mg or 750 mg of tremelimumab during one of the run-in cohorts, a lower dose level can be used in the main study. In addition, after completion of R3A and continuation in the main study phase, a control arm (Arm C) will be initiated where patients will be treated with tremelimumab monotherapy (without paclitaxel).

If no unexpected toxicity has occurred within 60 days after initiation of treatment of the 3rd patient of R3B, enrollment for run-in cohort R4 will begin in a similar fashion as described for the earlier run-in cohorts. Expansion arms A and C will be paused while this cohort is enrolling. If no unexpected toxicity has occurred within 60 days after initiation of treatment of the 3rd patient of R4, enrollment for arm R4 will be continued into the main study phase (as Arm B). If unacceptable toxicity is observed at 300 mg of tremelimumab in combination with 1500mg durvalumab, arm B, combining paclitaxel, tremelimumab and durvalumab, will be discontinued.

Main study:

Arm A:

* paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
* tremelimumab 750 mg on day 1 of cycles 2-6 and then every 12 weeks until week 45

Arm B:

* paclitaxel 70 mg/m2 on day 1, 8, 15 of cycles 1-6
* tremelimumab 300 mg once on day 1 of cycle 2
* durvalumab 1500 mg on day 1 of cycles 2-12, every four weeks (until week 49)

Arm C (control arm):

• tremelimumab 750 mg on day 1 of cycles 1-5 and then every 12 weeks until week 41

Enrollment will be halted when 12 patients are enrolled in each arm; this will include patients treated in R3 and R4 at the dose level used in the main study. These patients will be included in the efficacy analysis.

After the last patient has had the second evaluation scan, the Objective Response Rate (ORR) of each treatment arm will be evaluated. If one or more of the experimental arms has ≥2 responses, the study team will discuss continuation of one of the experimental arms to n=20 with the IDMC. In case 2 responses are seen in one of the arms prior to the second evaluation scan of the last patient, a decision on expansion of that arm may be recommended earlier.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, European Union [EU] Data Privacy Directive) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Patients with histologically or cytologically documented metastatic or irresectable (i.e. T4b, N1-3 and/or M1a/b) urothelial cell carcinoma (including renal pelvis, ureters, urinary bladder, and urethra).
3. Patients ineligible for cisplatin-based chemotherapy OR previous treatment with platinum-based chemotherapy, either in the neo-adjuvant setting or in any other setting. This is defined as progression on or after at least 2 cycles of platinum-based chemotherapy (e.g. MVAC, cisplatin/gemcitabine, carpoblatin/gemcitabine). Patients who had to stop platinum-based therapy because of toxicity after at least 2 cycles are eligible if progressive disease has been confirmed.
4. Previous treatment with anti-PD(L)1 immunotherapy. The following conditions apply for inclusion:

   1. Must not have experienced a toxicity that led to permanent discontinuation of prior anti-PD(L)1 immunotherapy;
   2. All treatment-related AEs while receiving prior anti-PD(L)1 immunotherapy must have completely resolved or resolved to baseline prior to screening for this study;
   3. Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior anti-PD(L)1 immunotherapy;
   4. Patients with endocrine AE of ≤Grade 2 are permitted to enroll if the AEs are stably maintained on appropriate replacement therapy and are asymptomatic;
   5. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of >10 mg prednisone or equivalent per day;
5. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have a Revised Clinical Study Protocol short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and that is suitable for accurate repeated measurements as per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) guidelines.
6. Age >18 years at time of study entry.
7. World Health Organisation (WHO) performance status of 0 or 1.
8. Body weight >30kg.
9. Adequate normal organ and marrow function as defined below:

   1. Haemoglobin ≥9.0 g/dL = 5.6 mmol/L;
   2. Absolute neutrophil count (ANC) ≥1.5 x 109/L;
   3. Platelet count ≥100 x 109/L;
   4. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). (Does not apply to patients with confirmed Gilbert's syndrome, who will be allowed only in consultation with the treating physician);
   5. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN;
   6. Measured creatinine clearance (CL) >30 mL/min or Calculated creatinine clearance CL>30 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal in case of amenorrhoeu for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal in case of amenorrhea for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy);
    * Women ≥50 years of age would be considered post-menopausal in case of amenorrhea for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy);
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
12. Must have a life expectancy of at least 12 weeks

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Participation in another clinical study with an investigational product during the last 4 weeks.
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
4. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) ≤28 days prior to the first dose of study drug.
5. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician;
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician;
   * Toxicity caused by treatment with anti-PD(L)1 should return to baseline, except for endocrine toxicity on a stable dose of replacement therapy.
6. Any concurrent chemotherapy, investigational product (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
7. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
8. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
9. History of allogenic organ transplantation.
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia;
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement;
    * Any chronic skin condition that does not require systemic therapy. Psoriasis, if not treated by immunesuppressants, is allowed;
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician;
    * Patients with celiac disease controlled by diet alone.
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
12. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of IP and of low potential risk for recurrence;
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease;
    * Adequately treated carcinoma in situ without evidence of disease;
    * Curatively treated localized prostate cancer without PSA recurrence.
13. History of leptomeningeal carcinomatosis.
14. Brain metastases or spinal cord compression, unless radiographically stable, defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression. In addition, any neurologic symptoms that developed either as a result of the brain metastases or treatment thereof must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤10mg/day of prednisone or its equivalent for at least 14 days prior to the start of treatment.. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry.
15. History of active primary immunodeficiency.
16. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection);
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent;
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
19. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of tremelimumab, durvalumab, or durvalumab + tremelimumab combination therapy.
20. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
21. Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
22. Previous treatment with anti-CTLA-4 immunotherapy.
23. Known allergy or hypersensitivity to IP or any excipient. Procedures for withdrawal of incorrectly enrolled patients are presented in Section 4.3 of the clinical protocol. If a patient withdraws from participation in the study, then that specific enrollment/randomization code cannot be reused. Withdrawn patients will not be replaced.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR), defined as the proportion of participants whose confirmed best overall response is either a PR or CR after treatment with paclitaxel and a high dose of tremelimumab based upon the RECIST v1.1 guidelines. | Final ORR will be determined after the confirmatory scan of the last patient, which is scheduled up to 21 weeks after start of treatment of the final patient
  Tumor evaluation will take place using CT-Chest and abdomen, based on the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) guidelines. The first evaluation will take place 12 weeks after initiating treatment. After this initial scan, tumor evaluation will take place every 8 weeks for the first year. After the first year, tumor evaluation will be done every 12 weeks.
Overall response rate (ORR), defined as the proportion of participants whose confirmed best overall response is either a PR or CR after treatment with paclitaxel, tremelimumab and durvalumab based upon the RECIST v1.1 guidelines. | Final ORR will be determined after the confirmatory scan of the last patient, which is scheduled up to 21 weeks after start of treatment of the final patient
  Tumor evaluation will take place using CT-Chest and abdomen, based on the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) guidelines. The first evaluation will take place 12 weeks after initiating treatment. After this initial scan, tumor evaluation will take place every 8 weeks for the first year. After the first year, tumor evaluation will be done every 12 weeks.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Overall therapeutic safety will be determined 90 days after the last patient has received the last treatment dose
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Overall survival (OS) in months for each of the treatment strategies. | OS data will be collected up to 2 years after inclusion of the final patient
  survival data will be collected every 6 months after the last study visit for each participant.
Progression-free survival (PFS) in months for each of the treatment strategies | PFS data will be collected up to 2 years after inclusion of the final patient
  survival data will be collected every 6 months after the last study visit for each participant.
Duration of response in months for each of the treatment strategies | DOR data will be collected up to 2 years after inclusion of the final patient
  survival data will be collected every 6 months after the last study visit for each participant.

OTHER OUTCOMES:
Determine the effects of paclitaxel +/- tremelimumab +/- durvalumab on T-cell infiltration in the tumor-immune micro-environment (TME) when comparing baseline vs on-treatment tumor biopsies. | Tissues and samples will be collected up to 2 years after inclusion of the final patient
  CD8+ T-cell infiltration has shown to correlate with response to checkpoint blockade therapy. Baseline versus on-treatment biopsies will be compared to determine whether CD8+ T-cell infiltration correlates with response to therapy and clinical efficacy parameters. CD8+ T-cell infiltration will be determined based on CD8+ IHC stainings and multiplex immunofluorescence.
Obtain a comprehensive overview of changes in the tumor micro-environment upon treatment with paclitaxel +/- tremelimumab +/- durvalumab comparing baseline and on-treatment biopsies. | Tissues and samples will be collected up to 2 years after inclusion of the final patient
  Apart from CD8+ T-cell infiltration, few markers have been identified that play a significant prognostic or predictive role in bladder cancer. An overview of the tumor micro-environment (TME) will be created using multiplex immunofluorescence and RNA expression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel MS van der Heijden, MD, PhD, Principal Investigator — NKI-AvL
Locations (1):
- Antoni van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands